CLINICAL TRIAL: NCT01737905
Title: Evaluation of Efficacy and Safety for Single Dose of E004 in Children With Asthma (A Randomized, Double-Blind, Placebo-Controlled, Crossover, Single Dose Study in 4 - 11 Year Old Children With Asthma)
Brief Title: Evaluation of Efficacy and Safety for Single Dose of E004 in Children With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amphastar Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: API-E004-CL-D2
Record Dates: First submitted 2012-11-20; First posted 2012-11-30 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-02

CONDITIONS: Asthma
Keywords: Asthma; Safety; Efficacy; Epinephrine; Bronchodilator; Metered dose inhaler
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm T (Experimental): Experimental arm utilizing Epinephrine HFA-MDI (E004)
  Interventions: Drug: Epinephrine HFA-MDI (E004)
- Arm P (Placebo Comparator): Placebo comparator arm utilizing Placebo-HFA
  Interventions: Drug: Placebo-HFA

INTERVENTIONS:
Drug: Epinephrine HFA-MDI (E004) — Single dose 125 mcg/inhalation, 2 inhalations
  Arms: Arm T
Drug: Placebo-HFA — Single dose 0 mcg/inhalation, 2 inhalations
  Arms: Arm P

SUMMARY:
This is a multi-center, randomized, double-blinded, placebo-controlled, crossover, single dose study in 24 pediatric patients (4-11 years old) with asthma.

The entire study consists of (i) a Screening Visit and (ii) a Study Period with two (2) Study Visits. All study subjects must be properly consented, under adult supervision, and screened against the inclusion and exclusion criteria, at the Screening Visit.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, placebo-controlled, crossover, single dose study to be conducted in pediatric patients (4 - 11 years) with asthma.

The main features of the study design are:

The entire study consists of a Screening Visit, and a Study Period consisting of two (2) crossover Study Visits separated by a 2 to 14-day interval. All study subjects must be properly consented, under adult supervision, and screened against the inclusion and exclusion criteria at the Screening Visit and confirmed for enrollment on Visit 1. Efficacy and safety evaluations of E004 are conducted at each Study Visit.

This study employs two (2) double-blinded treatment arms as outlined in Table 2. A double-blinded design will be applied to E004 (Arm T) and Placebo-HFA (Arm P) since they are identical in all physical attributes and share a comparable formulation.

The enrolled subjects will be randomized into two sequences (as follows) to participate in two (2) crossover Study Visits with a 2 - 14 day interval between visits. Randomization is achieved using a ratio of 1:1.

Use E004 (T) and Placebo (P) in Visits 1 and 2, respectively or use Placebo (P) and E004 (T) in Visits 1 and 2, respectively

Subjects will be trained at the screening visit and each Study Visit for the correct dosing and spirometry methods. Under the supervision of dosing monitor, subjects will self-administer two (2) inhalations of the randomized study treatment, with a ~1 min interval at each Study Visit.

For the Screening and Study Visits, the subjects will be required to be at the site for a 30 minute "resting period". This resting period is designed to maintain a stable and consistent physical status of the subjects prior to the start of the baseline FEV1 procedures. For the Screening Visit, this period will begin upon subject arrival. For the Study Visits, the period will begin at the end of the option breakfast (or upon arrival if the breakfast is declined).

For each Study Visit, subjects will need to arrive at the study site early enough to complete all necessary baseline evaluations. The study site will provide an optional breakfast but it must be eaten at least 30 minutes prior to the pre-dose baseline FEV1 measurements. The optional breakfast will be light, and contain no added sugar. If the subjects decline the breakfast (i.e. they have already eaten a light breakfast prior to arriving), they are required to remain at the site for at least 30 minutes prior to the start of the Baseline FEV1 measurements, in order to maintain a stable physical status.

Baseline vital signs and safety evaluations will be taken prior to the pre-dose baseline FEV1 measurement. These can be performed during the 30 minute "resting period". Efficacy of the treatments at each visit will be evaluated based on spirometric measurements of serial FEV1 determined at the Pre-dose Baseline, and the seven (7) serial Post-dose FEV1 responses at 5, 30, 60, 120, 150, 180) and 240 minutes.

This study will be conducted with a double-blinded technique. This means neither the subject nor the site staff will be aware of the identity of the treatment arm since both study treatments are in identical looking containers.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy male, and premenarchal female, children ages 4 - 11 years upon Screening.
* With documented asthma, requiring inhaled epinephrine or β2-agonist treatment, with or without concurrent anti-inflammatory therapies including orally inhaled corticosteroids, for at least 6-months prior to Screening.
* Being capable of performing spirometry for FEV1 measurements.
* Satisfying criteria of asthma stability, defined as no significant changes in asthma therapy (with the exception of switching LABA to SABA, adjustment of ICor SABA, etc, per investigator discretion) and no asthma-related hospitalization or emergency room visits, within 4 weeks prior to Screening.
* Can tolerate withholding treatment with inhaled bronchodilators and other allowed medications for the minimum washout periods indicated in Appendix II prior to the Screening Baseline FEV1 testing.
* Demonstrating a Mean Screening Baseline FEV1 (MSBF) that is 50.0% - 90% of Polgar predicted normal value.
* Demonstrating an Airway Reversibility, i.e., FEV1 values ≥12% increase based upon volume compared with MSBF, within 30 min after 2 inhalations (440 mcg, epinephrine base) of previously marketed Epinephrine CFC-MDI, labeled "For Investigational Use Only". There will be up to 5 reversibility time points, each with up to 5 maneuvers that can be conducted anytime within 30 min post-dose.
* Demonstrating satisfactory techniques in the use of a metered-dose inhaler (MDI).
* Has been properly consented to participate in this study.

Exclusion Criteria:

* Any current or past medical conditions that, per investigator discretion, might significantly affect pharmacodynamic responses to the study drugs, such as significant systemic or respiratory diseases (e.g., cystic fibrosis, bronchiectasis, active tuberculosis, emphysema, nonreversible pulmonary diseases), other than asthma.
* Concurrent clinically significant cardiovascular, hematological, renal, neurologic, hepatic, endocrine, psychiatric, or malignant diseases.
* Known intolerance or hypersensitivity to any component of the study drugs (i.e., Epinephrine, HFA-134a, CFC-12, CFC-114, polysorbate-80, thymol, ethanol, ascorbic acid, nitric acid, and hydrochloric acid), as well as the rescue Albuterol HFA inhalers (i.e., Albuterol, HFA-134a, ethanol, and oleic acid).
* Recent infection of the upper respiratory tract (within 2 weeks), or lower respiratory tract (within 4 weeks), before screening.
* Use of prohibited medications per Appendix II.
* Having been on other investigational drug/device studies in the last 30 days prior to screening.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Bronchodilator effect | up to 30 min pre-dose, postdose up to 3 hours
  Bronchodilator effect expressed as AUC of FEV1's relative change from the same day baseline (pre-dose) versus time up to 3 hours, defined as AUC(0-3) of change in FEV1%. The difference of primary endpoints of E004 and Placebo will be evaluated statistically.

SECONDARY OUTCOMES:
AUC analysis | up to 30 min pre-dose, postdose up to 3 hours
  The comparative analysis of AUC of FEV1 versus time
Evaluation of FEV1 volume changes | up to 30 min pre-dose, postdose up to 3 hours
  Evaluation of AUC(0-3) and AUC(0-4) of FEV1 volume changes (AUC of ΔFEV1)
Change in FEV1 | up to 30 min pre-dose, postdose up to 3 hours
  Evaluation of Maximum of change in FEV1% (Fmax)
Time response | up to 30 min pre-dose, postdose up to 3 hours
  Evaluation of time response curves of change in FEV1 and FEV1%
Time to onset of bronchodilator effect | up to 30 min pre-dose, postdose up to 3 hours
  Determination of time to onset of bronchodilator effect (Tonset), determined by the time point (within 60 minutes) where FEV1 first reaches greater than or equal to 12% above Same-Day Pre-dose Baseline
Time to peak FEV1 effect | up to 30 min pre-dose, postdose up to 3 hours
  The time to peak FEV1 effect (Tmax), defined as the time of Fmax
Duration of efficacy | up to 30 min pre-dose, postdose up to 3 hours
  Evaluation of duration of efficacy (Tduration), defined as the total length of time when the change in FEV1% reaches and stays greater than or equal to 12% above Same-Day Pre-dose Baseline
Percentage of positive responders | up to 30 min pre-dose, postdose up to 3 hours
  Evaluation of percentage of positive responders (R%), including all subjects whose Fmax reaches more than or equal to 12% above Same-Day Pre-dose Baseline
Vital Signs | Screening Visit: baseline up to 30 min predose and 30 min post dose; Visits 1-2: Baseline upt o 30 min predose and 3, 20, 60, and 240 min post-dose
  Vital signs (SBP/DBP, and heart rate) will be monitored at the Screening Visit and at Study Visits 1 and 2
12-lead ECG (Routine and QT/QTc) | Screening Visit: baseline up to 30 min predose and 30 min post dose; Visits 1-2: Baseline upt o 30 min predose and 3, 20, and 60 min post-dose
  A 12-lead ECG (Routine and QT/QTc) will be recorded at Screening Visit and at the Study Visits 1 and 2
Lab Tests | prior to first dose
  Lab tests for CBC, blood chemistry panel (8-hr fasted), and urinalysis will be performed at screening
Albuterol HFA Usage | up to 30 min predose
  Albuterol HFA usage for rescue relief of acute asthma symptoms will be recorded at each visit
Concomitant Medications | up to 30 min predose
  Concomitant medications will be reviewed and recorded
Adverse Events | predose and up to 3 hours postdose
  All Adverse Events/side effects will be recorded and assessed

CONTACTS AND LOCATIONS:
Overall Officials: Selina Su, MPH, Study Director — Amphastar Pharmaceuticals, Inc.
Locations (6):
- United States (6):
  - West Coast Clinical Trials Global, Cypress, California
  - The Clinical Research Institute of Southern Oregn, PC, Medford, Oregon
  - Transitional Clinical Research, Inc. Allergy Associates Research Center, Portland, Oregon
  - Western Sky Medical, El Paso, Texas
  - Sylvana Research Assocaites, San Antonio, Texas
  - ASTHMA, Inc. Clinical Research Center, Seattle, Washington

REFERENCES:
- [Background] Pinnas JL, Schachtel BP, Chen TM, Roseberry HR, Thoden WR. Inhaled epinephrine and oral theophylline-ephedrine in the treatment of asthma. J Clin Pharmacol. 1991 Mar;31(3):243-7. doi: 10.1002/j.1552-4604.1991.tb04969.x. PMID 2019665
- [Background] Hendeles L, Marshik PL, Ahrens R, Kifle Y, Shuster J. Response to nonprescription epinephrine inhaler during nocturnal asthma. Ann Allergy Asthma Immunol. 2005 Dec;95(6):530-4. doi: 10.1016/S1081-1206(10)61014-9. PMID 16400891
- [Background] Warren JB, Doble N, Dalton N, Ewan PW. Systemic absorption of inhaled epinephrine. Clin Pharmacol Ther. 1986 Dec;40(6):673-8. doi: 10.1038/clpt.1986.243. PMID 3780129
- [Background] Cripps A, Riebe M, Schulze M, Woodhouse R. Pharmaceutical transition to non-CFC pressurized metered dose inhalers. Respir Med. 2000 Jun;94 Suppl B:S3-9. PMID 10919679
- [Background] Dickinson BD, Altman RD, Deitchman SD, Champion HC. Safety of over-the-counter inhalers for asthma: report of the council on scientific affairs. Chest. 2000 Aug;118(2):522-6. doi: 10.1378/chest.118.2.522. PMID 10936150
- [Background] Simons FE, Gu X, Johnston LM, Simons KJ. Can epinephrine inhalations be substituted for epinephrine injection in children at risk for systemic anaphylaxis? Pediatrics. 2000 Nov;106(5):1040-4. doi: 10.1542/peds.106.5.1040. PMID 11061773
- [Background] Hankinson JL, Odencrantz JR, Fedan KB. Spirometric reference values from a sample of the general U.S. population. Am J Respir Crit Care Med. 1999 Jan;159(1):179-87. doi: 10.1164/ajrccm.159.1.9712108. PMID 9872837